CLINICAL TRIAL: NCT06348212
Title: Effect of Probiotic Strain Lactobacillus Paracasei PS23 on Brain Fog in People With Long COVID
Acronym: COVID-19
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, Ching-Liang Lu, director of endoscopy center, Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-11-008C
Record Dates: First submitted 2024-03-18; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Long COVID; Brain Fog; Cognitive Change
Keywords: Probiotics; EEG; Gut brain axis
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Mental Fatigue | interventions — microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomization were performed by the provider of probiotic and placebo. The participant will never know their group. The study Investigator and Outcome assessor will not know the groups of participants until they finish recruiting and data processing.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental): They are given probiotic capsules of Lactobacillus paracasei PS23. Each capsule contains 100 mg of probiotic powder(10,000,000,000 CFU) Subjects should take two capsules per day for two months
  Interventions: Dietary Supplement: Lactobacillus paracasei PS23
- Placebo group (Placebo Comparator): They are given probiotic capsules of microcrystalline cellulose. Subjects should take two capsules per day for two months
  Interventions: Dietary Supplement: microcrystalline cellulose

INTERVENTIONS:
Dietary Supplement: Lactobacillus paracasei PS23 — 2 caps daily use
  Arms: Probiotic group
Dietary Supplement: microcrystalline cellulose — 2 caps daily use
  Arms: Placebo group

SUMMARY:
The goal of this clinical trial is to test whether the intervention of probiotics supplement can improve symptoms of long covid syndrome.

Participants will be given probiotics or placebo capsules for two month. Symptom questionnaires, cognitive function, eeg and fecal sample are recorded/collected before and after the supplement.

Researchers will compare the probiotic group and the placebo to see if probiotic supplement really make differences.

DETAILED DESCRIPTION:
After the pandemic of covid-19, people found out that not only does it cause acute respiratory system symptoms, but it also affect many other systems even long after the acute symptoms have resolved, which is named the Long Covid Syndrome. Studies have shown that the gut microbiota of those suffering from long covid syndrome differ from that of healthy people and those who recovered from covid without getting long covid syndrome, which implied the possibility of probiotic supplement being an effective treatment to long covid. This double-blind parallel randomized control trail plans to supply participants with probiotics or placebo fortwo months. Symptom questionnaires, cognitive function, eeg and fecal sample will be recorded/collected before and after the supplement. Researchers will compare the two groups to see if they differ in the above measure and to see if the differences in symptoms and cognitive functions change correlate with gut microbiota change and fecal metabolite change.

ELIGIBILITY:
Inclusion Criteria:

* 20 to 80 year old
* had been infected by SARS-CoV-2
* Stable vital signs
* Have brain fog conplaint
* MoCA<30 at baseline

Exclusion Criteria:

* refuse to join the study or refuse to sign the Informed Consent Form
* have other neurological disease that may affect cognitive function, such as Parkinson disease, Seizure, etc.
* have other gastrointestinal disease that may affect cognitive function, including tumors.
* severe hearing loss or visual loss that may hinder cognitive function tests
* Taken anti-seizure drug in 7 days.
* Already taking probiotics supplement regularly
* Taken antibiotics in two weeks
* taking stool softener or laxative regularly
* have valvular heart disease
* have congenital or acquired immunodeficiency or is under iimmunosuppressant therapy
* Pregnant or plans to be pregnant
* BMI>30
* Have been performed severe gastrointestinal surgery(s)
* Severe liver, kidney, cardiovascular, hematologic or metabolic disorder
* In critical condition

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Long covid related symptoms | baseline and two months after probiotic/placebo supplement
  A list of symptoms related to long covid including cough, fatigue. brain fog etc.
Hospital Anxiety and Depression Scale | baseline and two months after probiotic/placebo supplement
  A measurement of the degree of depression and anxiety, with 7 questions each and 0-3 points for each question. Two scores ranging from 0-21 will be calculated, with higher points meaning more severe depression or anxiety.
The Pittsburgh sleep quality index | baseline and two months after probiotic/placebo supplement
  A measurement of the degree of sleep disturbance/disorder. The score ranges from 0-21, with higher points meaning more severe sleep problem.
Fatigue Severity Scale | baseline and two months after probiotic/placebo supplement
  A measurement of the degree of fatigue, with score ranging from 7-49 and higher points meaning more severe fatigue.
GI symptoms | baseline and two months after probiotic/placebo supplement
  Rome Criteria Questionnaire in functional UGI disease and Rome Criteria Questionnaire in IBS are included in the questionnaire are measured to see if probiotic/placebo supplement results in adverse gi events or a change of bowel habits.
Cognitive function-Digit symbol substitution test | baseline and two months after probiotic/placebo supplement
  a list of paired numbers and symbols are given to participants, and they are ask to match symbols to numbers accordingly. The number of question they answer within 90 second will be recorded.
Cognitive function-The Montreal Cognitive Assessment(MoCA) | baseline and two months after probiotic/placebo supplement
  Score ranging from 0-30, with higher meaning better cognitive function
Cognitive function-Color Trails making Test | baseline and two months after probiotic/placebo supplement
  The test is composed of two parts, easy and hard. The time taken to finish the two parts are recorded
Cognitive function-Cogstate Brief Battery (CBB) | baseline and two months after probiotic/placebo supplement
  A cognitive test on ipad.
EEG | baseline and two months after probiotic/placebo supplement
  2 minutes of resting-state eye-open eeg were recored. After a brief rest, a working memory task will be repeated for 12 times.
  In the task, subjects will be shown balls in a 5*5 chart, the location of which They are asked to remember. 6 second later, they are shown another ball, and they will be asked if the location of the newly shown ball are identical with any of the originally shown balls.
Gut microbiota | baseline and two months after probiotic/placebo supplement
  Subjects will be asked to collect their fecal sample and the bacterial DNA/RNA will be extracted and analyzed.
Fecal metabolite | baseline and two months after probiotic/placebo supplement
  Subjects will be asked to collect their fecal sample and the SCFAs in the sample will be measured.

IPD SHARING:
Plan to Share IPD: No